CLINICAL TRIAL: NCT01294241
Title: Open, Prospective, Controlled Case Series Documentation to Compare Intra-individually the Efficacy and Tolerance of Sericare® Versus Non-adhesive Wound Dressing Alone in Accelerating the Epithelialization of Skin Lesions of Patients With Epidermolysis Bullosa Hereditaria
Brief Title: Oleogel-S10 in Wound Healing of Inherited Epidermolysis Bullosa (BEB-10)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Birken AG (Industry)
Responsible Party: Sponsor
Organization: Amryt Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BEB-10
Record Dates: First submitted 2010-10-27; First posted 2011-02-11 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-05

CONDITIONS: Inherited Epidermolysis Bullosa
Keywords: Epidermolysis bullosa; Wound healing; Epithelialization
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded comparison of wound photo series by two independent experts
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oleogel-S10 (Experimental): The eligible wound (half) was topically treated with Oleogel-S10 and covered with a non-adhesive wound dressing (Mepilex®) on Day 0. Wound dressings were changed about every 24 to 48 hours until discharge from hospital or until the end of treatment at Day 14 in 'recent wounds' or Day 28 in 'chronic wounds'.
  Interventions: Drug: Oleogel-S10; Device: Mepilex® soft silicone faced polyurethane foam dressing
- Non-adhesive wound dressing (Other): Mepilex® soft silicone faced polyurethane foam dressing was used as non-active comparator. The eligible wound (half) was covered with Mepilex® as control on Day 0. Wound dressings were changed about every 24 to 48 hours until discharge from hospital or until the end of treatment at Day 14 in 'recent wounds' or Day 28 in 'chronic wounds'.
  Interventions: Device: Mepilex® soft silicone faced polyurethane foam dressing

INTERVENTIONS:
Drug: Oleogel-S10 — 1 cm or 125 µL or 115 mg Oleogel-S10 per cm2 wound area (corresponds to thickness of approximately 1 mm or 0.04 inch) every 24 to 48 hours until discharge from hospital or until the end of treatment at Day 14 in 'recent wounds' or Day 28 in 'chronic wounds'.
  Other Names: Sericare®
  Arms: Oleogel-S10
Device: Mepilex® soft silicone faced polyurethane foam dressing — Mepilex® soft silicone faced polyurethane foam dressing was changed about every 24 to 48 hours until discharge from hospital or until the end of treatment at Day 14 in 'recent wounds' or Day 28 in 'chronic wounds'.
  Other Names: Cutaneous patch

SUMMARY:
The purpose of this study was to compare intra-individually the reepithelialization of skin lesion(s) in inherited Epidermolysis bullosa (either 1 wound ≥10 cm2 and ≤200 cm2 in size divided in 2 equal halves or 2 comparable wounds of ≥5 cm2 each) treated with Oleogel-S10 and non-adhesive wound dressing versus non-adhesive wound dressing only.

DETAILED DESCRIPTION:
This study was designed as an open-label, prospective, controlled, blindly evaluated, monocentric phase II case series documentation in patients with inherited Epidermolysis bullosa (EB). The investigator either identified 1 EB wound ≥10 cm2 and ≤200 cm2 in size and divided it into 2 halves or selected 2 comparable wounds of ≥5 cm2 each. One (half of the) EB wound was treated with Oleogel-S10 and non-adhesive wound dressing. The other wound (half) was covered with a non-adhesive wound dressing only (Mepilex®) as control. Wound dressings were changed about every 24 to 48 hours until discharge from hospital or until the end of treatment at Day 14 in 'recent wounds' or Day 28 in 'chronic wounds'. This was an open-label study. The investigator, the participant, and the sponsor knew the identity of the treatment. Two independent experts were blind to treatment and assessed efficacy based on chronological series of cropped and coded photographs by wound (half) that were taken before start of treatment, during wound dressing changes and at the end of treatment on Day 14/Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 1-95 years
2. Patient and/or his/her legal representative was informed, read and understood the patient information/informed consent form and gave written informed consent
3. Patients with inherited EB with at least 1 skin lesion between 10 cm2 and 200 cm2 (alternatively 2 comparable lesions of at least 5 cm2 each)
4. Patient and/or his/her legal representative was able and willing to follow study procedures and instructions including the following:

   1. Application of Oleogel-S10 on (1 half of) the wound at every wound dressing change
   2. Regular visits during the treatment period (14 days in 'recent wounds' to 28 days in 'chronic wounds')
5. Negative pregnancy test in women of childbearing potential within 7 days before start of treatment
6. Women of childbearing potential agreed to use an effective method of contraception (Pearl Index < 1, e.g. hormonal contraception including the combined oral contraceptive pill, the transdermal patch, and the contraceptive vaginal ring, intrauterine devices or sterilization) during treatment and for at least 6 months thereafter
7. Men of procreative capacity agreed to use an effective method of contraception during treatment and for at least 6 months thereafter

Exclusion Criteria:

1. Systemic treatment with steroids during the last 30 days
2. Uncontrolled diabetes mellitus or diabetic ulcers
3. Diseases or conditions that could, in the opinion of the investigator, interfere with the assessment of safety, tolerance or efficacy
4. Skin disorders adversely affecting wound healing or involving the areas eligible for study treatment
5. Hypersensitivity to the trial medication or surgical dressings to be used
6. Multiple allergic disorders
7. Administration of investigational drugs within 3 months before screening
8. Investigations or changes in management for an existing medical condition
9. Low probability to complete the study per protocol for whatever reason

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Schwieger-Briel, MD, Principal Investigator — University Medical Center Freiburg
Locations (1):
- EB Center at the Department of Dermatology, University Medical Center, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 03 Nov 2010 to 14 Jun 2011 at 1 center (University Medical Center Freiburg) in 1 country (Germany).
Pre-assignment Details: 12 wounds in 10 participants (2 cycles of treatment in 2 participants) were treated with study medication. The reepithelialization was compared intra-individually in either 2 halves of an Epidermolysis bullosa (EB) wound ≥10 cm2 and ≤200 cm2 in size or in 2 EB wounds ≥5 cm2 in size, i.e. the total number of participants was 10 in the overall study.
Units Other Than Participants: Wounds
Groups:
- All Study Participants: One (half of an) EB wound ≥10 cm2 and ≤200 cm2 in size or 1 EB wound ≥5 cm2 in size was treated with Oleogel-S10 and non-adhesive wound dressing. The other wound (half) was covered with a non-adhesive wound dressing only (Mepilex®) as control (intra-individual comparison).
Period: Overall Study
Arm/Group | All Study Participants
Started | 10; 12 Wounds
Completed | 10; 12 Wounds
Not Completed | 0; 0 Wounds

BASELINE CHARACTERISTICS:
Population: As 2 participants received 2 cycles of treatment each, 12 wounds were treated with study medication.
Units Other Than Participants: Wounds
Groups:
- All Study Participants: One (half of an) EB wound ≥10 cm2 and ≤200 cm2 in size or 1 EB wound ≥5 cm2 in size was treated with Oleogel-S10 and non-adhesive wound dressing. The other wound (half) was covered with a non-adhesive wound dressing only (Mepilex®) as control.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Number analyzed (Wounds) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 20 [6 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  Germany | 10

OUTCOME MEASURES:

1. Primary Outcome: Intra-individual Difference in Reepithelialization of Wound (Halves) at Day 14 in 'Recent Wounds' or Day 28 in 'Chronic Wounds'
Description: The primary end point was the progress of reepithelialization from baseline to either Day 14 ('recent wounds') or Day 28 ('chronic wounds') of the EB wound (half) treated with Oleogel-S10 and non-adhesive wound dressing (Mepilex®) intra-individually compared to the other wound (half) covered with non-adhesive wound dressing only (intra-individual comparison). Two independent experts were blind to treatment and assessed efficacy based on chronological series of cropped and coded photographs by wound (half) that were taken before start of treatment, during wound dressing changes and at the end of treatment on Day 14/Day 28. They evaluated each series and decided whether 1 wound (half) reepithelialized faster than the other ('winner'), or whether there was no difference in reepithelialization.
Time Frame: 14 days for 'recent wounds', 28 days for 'chronic wounds'
Population: 12 wounds in 10 participants (intra-individual comparison, 2 cycles of treatment in 2 participants) were evaluated by assessors that were blind to treatment. 'Undecided' wounds that were either evaluated controversially (n=2) or as being equal (n=2) were excluded from the analysis of the primary efficacy variable.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Groups:
- All Study Participants: Intra-individual comparison of two treatments: One half of an EB wound ≥10 cm2 and ≤200 cm2 in size or 1 EB wound ≥5 cm2 in size was treated with Oleogel-S10 and non-adhesive wound dressing. The other wound (half) was covered with a non-adhesive wound dressing only (Mepilex®) as standard of care control.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Number analyzed (Wounds) | 8
Wounds
  Faster healing of wound treated with Oleogel-S10 | 8
  Faster healing of wound treated with dressing | 0
Statistical Analysis 1: Comparison: All Study Participants; The intra-individual difference in reepithelialization of wound (halves) was tested using a two-sided exact binomial test. The test was performed at a significance level of 5% for the null-hypothesis of no difference δ = 0 against the hypotheses δ ≠ 0: H0: δ = 0 H1: δ ≠ 0; Test type: Superiority or Other; p = 0.008, Two-sided exact binomial test — Post-hoc superiority analysis: Wounds that were either evaluated controversially (n=2) or as being equal (n=2) were excluded from the analysis of the primary efficacy variable

2. Secondary Outcome: Percentage of Wound Epithelialization at Day 7±1
Description: The secondary endpoint was the intra-individual difference in median percentage of wound epithelialization at Day 7±1. Sizes of wound areas were measured using a digital wound evaluation program from the EB Center at the Department of Dermatology, University Medical Center Freiburg.
Time Frame: Day 7±1
Population: As 2 participants received 2 cycles of treatment each, 12 wounds were treated with study medication.
Measure: Median (Full Range); unit: Percentage of wound epithelialization
Units Other Than Participants: Wounds/wound halves
Groups:
- Oleogel-S10 and Non-adhesive Wound Dressing: One half of an EB wound ≥10 cm2 and ≤200 cm2 in size or 1 EB wound ≥5 cm2 in size was treated with Oleogel-S10 and non-adhesive wound dressing.
- Non-adhesive Wound Dressing Only: The other half of an EB wound ≥10 cm2 and ≤200 cm2 in size or 1 EB wound ≥5 cm2 in size was treated with non-adhesive wound Dressing only as control.
Arm/Group | Oleogel-S10 and Non-adhesive Wound Dressing | Non-adhesive Wound Dressing Only
Number analyzed (Participants) | 10 | 10
Number analyzed (Wounds/wound halves) | 12 | 12
Percentage of wound epithelialization | 69.7 [17.3 to 90.4] | 57.4 [10.0 to 81.3]
Statistical Analysis 1: Comparison: Oleogel-S10 and Non-adhesive Wound Dressing; The intra-individual difference in median percentage of wound epithelialization was tested using a two-sided Wilcoxon test; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney) — Post-hoc superiority analysis

3. Secondary Outcome: Percentage of Wound Epithelialization at Day 14±1
Description: The secondary endpoint was the intra-individual difference in median percentage of wound epithelialization at Day 14±1. Sizes of wound areas were measured using a digital wound evaluation program from the EB Center at the Department of Dermatology, University Medical Center Freiburg.
Time Frame: Day 14±1
Population: As 2 participants received 2 cycles of treatment each, 12 wounds were treated with study medication.
Measure: Median (Full Range); unit: Percentage of wound epithelialization
Units Other Than Participants: Wounds/wound halves
Arm/Group | Oleogel-S10 and Non-adhesive Wound Dressing | Non-adhesive Wound Dressing Only
Number analyzed (Participants) | 10 | 10
Number analyzed (Wounds/wound halves) | 12 | 12
Percentage of wound epithelialization | 87.7 [2.7 to 100.0] | 79.2 [0.0 to 98.3]
Statistical Analysis 1: Comparison: Oleogel-S10 and Non-adhesive Wound Dressing; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney) — Post-hoc superiority analysis

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from start of study treatment (Day 0) to completion of study treatment (Day 14/Day 28), i.e. for a period of up to 2 or 4 weeks.
Groups:
- Safety Population: All participants who received at least 1 dose of Oleogel-S10 were included in the safety population. All adverse events were reported for all study participants. Localized adverse events were not separately reported by intervention.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=10)
Wound area increased due to trauma/wound dressing change (Skin and subcutaneous tissue disorders) | 5 (9)
Wound infection (Skin and subcutaneous tissue disorders) | 1 (1)
Flu-like syndrome (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, subjects with dystrophic Epidermolysis bullosa only, difficult wound size analysis at fixed study days due to several episodes of re-trauma in both intervention and control wounds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No